CLINICAL TRIAL: NCT02255604
Title: Effect of Intralymphatic Immunotherapy at Basophil Response and Plasmacell Kinetic in Patients With Allergic Rhinitis.
Brief Title: Effect of Intralymphatic Immunotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ILIT
Record Dates: First submitted 2014-09-17; First posted 2014-10-02 (Estimated); Results first posted 2021-03-18 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2017-02

CONDITIONS: Allergy; Immune Tolerance; Injection Site Discomfort
Keywords: Allergic Rhinitis; Allergen immunotherapy
MeSH Terms: conditions — Hypersensitivity; Rhinitis, Allergic | interventions — Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- intralymphatic immune therapy (Active Comparator): Lymphnodes in the groin are identified with ultrasound. Under ultrasound guide they are injected with 0,1 ml of alk 225 Phleum Pratense 10,000 standard quantity units/ml.
  Patients receive 4 injection in total. 3 injection in the spring 2014 with one month interval and 1 injection in the spring 2015.
  Interventions: Drug: Alk (225) Phleum Pratense. 0.1 ml of 10,000 standard quantity units/ml.
- 3 intralymphatic immune therapy (Placebo Comparator): Lymphnodes in the groin are identified with ultrasound. Under ultrasound guide they are injected with 0,1 ml of alk 225 Phleum Pratense 10,000 standard quantity units/ml.
  Patients receive 3 injection in total. 3 injection in the spring 2014 with one month interval. In in the spring 2015 patients will have a placebo injection.
  Interventions: Drug: alk (225) Phleum Pratense. 0.1 ml of 10,000 standard quantity units/ml.
- no intralymphatic immune therapy (Sham Comparator): Lymphnodes in the groin are identified with ultrasound. Under ultrasound guide they are injected with 0,1 ml of isotone saline.
  Patients receive 4 injection in total. 3 injection in the spring 2014 with one month interval and 1 injection in the spring 2015. All injections are with isotone saline as placebo control.
  Interventions: Drug: 0.1 ml Isoton saline

INTERVENTIONS:
Drug: Alk (225) Phleum Pratense. 0.1 ml of 10,000 standard quantity units/ml. — 4
  Arms: intralymphatic immune therapy
Drug: alk (225) Phleum Pratense. 0.1 ml of 10,000 standard quantity units/ml. — 3 injection into a lymphnode
  Arms: 3 intralymphatic immune therapy
Drug: 0.1 ml Isoton saline — 4 injection into a lymphnode
  Arms: no intralymphatic immune therapy

SUMMARY:
The investigators want to investigate whether specific immunotherapy can be delivered directly into a lymph node. The investigators think that a direct introduction of allergen to the antigen presenting cells in the lymph node a give a strong immune response and that this can change the number of injections needed in allergen immunotherapy. The investigators do measurements of clinical effect and a variety of paraclinical test to see if the investigators can find af biomarker of successful specific immune therapy of grass allergy.

DETAILED DESCRIPTION:
Patients are injected with 3 or 4 doses of alk 225 Phleum Pratense 1000 standard quantity units/ml in a lymph node in the groin.

The investigators monitor clinical response and use of medication during the grass pollen season. SMS (Symptom and Medication Score) will be used.

The investigators count the number of immunoglobulin E grass producing plasma cells in blood one week after each injection. The investigators also do basophil activation tests, nasal provocation tests and titrated skin prick test to monitor effect.

Adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Allergic rhinitis to grass pollen, more than 3 mm reaction at skin prick test for grass, age between 18 and 40 years.

Exclusion Criteria:

* Uncontrolled asthma.
* Severe asthma with post bronchodilator test forced expiratory volume at 1 second less than 70% of expected.
* Severe co morbidity. Allergy to Fenol or Aluminium hydroxid.
* Any autoimmune diseases. Treatment with beta blocking medicine.
* Any heart diseases.
* Severe arterial hypertension. Kidney failure.
* Known malignancy. Known pregnancy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-08; Primary Completion 2015-09 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Søren Helbo SH Skaarup, MD, Principal Investigator — Lungemedicinsk forskningsafdeling. Aarhus University Hospital.
Locations (1):
- Lungemedicinsk Forskningsafdeling. Aarhus University Hospital, Aarhus, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Intralymphatic Immune Therapy: Lymphnodes in the groin are identified with ultrasound. Under ultrasound guide they are injected with 0,1 ml of alk 225 Phleum Pratense 10,000 standard quantity units/ml.
  Patients receive 4 injection in total. 3 injection in the spring 2014 with one month interval and 1 injection in the spring 2015.
  Alk (225) Phleum Pratense. 0.1 ml of 10,000 standard quantity units/ml.: 4
- 3 Intralymphatic Immune Therapy: Lymphnodes in the groin are identified with ultrasound. Under ultrasound guide they are injected with 0,1 ml of alk 225 Phleum Pratense 10,000 standard quantity units/ml.
  Patients receive 3 injection in total. 3 injection in the spring 2014 with one month interval. In in the spring 2015 patients will have a placebo injection.
  alk (225) Phleum Pratense. 0.1 ml of 10,000 standard quantity units/ml.: 3 injection into a lymphnode
- no Intralymphatic Immune Therapy: Lymphnodes in the groin are identified with ultrasound. Under ultrasound guide they are injected with 0,1 ml of isotone saline.
  Patients receive 4 injection in total. 3 injection in the spring 2014 with one month interval and 1 injection in the spring 2015. All injections are with isotone saline as placebo control.
  0.1 ml Isoton saline: 4 injection into a lymphnode
Period: Overall Study
Arm/Group | Intralymphatic Immune Therapy | 3 Intralymphatic Immune Therapy | no Intralymphatic Immune Therapy
Started | 12 | 12 | 12
Completed | 10 | 11 | 9
Not Completed | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intralymphatic Immune Therapy | 3 Intralymphatic Immune Therapy | no Intralymphatic Immune Therapy | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.67 (5.52) | 29.92 (6.80) | 30.58 (7.43) | 30.72 (6.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 5 | 17
  Male | 4 | 8 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in cSMS (Combined Symptom and Medication Score)
Description: cSMS, Combined symptom and medication score, during grass pollen season in three years follow up.
  Minimal score 0, Maximal score 18. Higher score means worse outcome.
  Scale:
  Itchy/red eys: 0-3, Runny eyes: 0-3, Itchy nose: 0-3, Runny nose: 0-3, Block nose: 0-3, Sneezes: 0-3. Topical antihistamine 1.5 points/1 point. Nasal corticosteroid: 1 point/2 points. Oral antihistamine: 6 points/1 point. Oral prednisolon 1.5 point /3 points.
  Elements are summed to a combined score. Different combination methods exists. EAACI recommends means, i.e. symptoms 0-3 plus medicationscore 0-3. This scoringsystem was applied in the last follow-up year.
Time Frame: 3 years
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intralymphatic Immune Therapy | 3 Intralymphatic Immune Therapy | no Intralymphatic Immune Therapy
Number analyzed (Participants) | 10 | 11 | 9
score on a scale | 2.6 [1.8 to 3.4] | 2.3 [1.5 to 3.0] | 4.5 [3 to 6]

2. Secondary Outcome: Change in Circulating Grass Specific Immunoglobulin E Producing Plasmacells
Time Frame: one week from vaccinations
Population: Due to technical flow-cytometry problem could analysis of circulating grass specific immunoglobulin E producing plasma cells not be performed.
Arm/Group | Intralymphatic Immune Therapy | 3 Intralymphatic Immune Therapy | no Intralymphatic Immune Therapy
Number analyzed (Participants) | 0 | 0 | 0

3. Other Pre Specified Outcome: Change in Basophil Sensitivity
Description: Flowcytometry based analysis of basophil cells reaction to allergen provocation.
Time Frame: 2 years
Population: Due to technical problems data was not recorded at all time points and results are missing.
Arm/Group | Intralymphatic Immune Therapy | 3 Intralymphatic Immune Therapy | no Intralymphatic Immune Therapy
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Intralymphatic Immune Therapy | 3 Intralymphatic Immune Therapy | no Intralymphatic Immune Therapy
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 7/12 | 5/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intralymphatic Immune Therapy (N=12) | 3 Intralymphatic Immune Therapy (N=12) | no Intralymphatic Immune Therapy (N=12)
Local reaction (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) | 0 (0) — Local swelling, edema and rubor at injection point
Headache (Immune system disorders) | 3 (3) | 0 (0) | 1 (1) — Headache, fatigue
anaphylaxis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) — anaphylaxis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No